CLINICAL TRIAL: NCT00309361
Title: A Phase 3, Multicenter, Randomized, Blinded, Controlled Study of NV-101 for Efficacy, Pharmacodynamics and Safety in Dental Patients Undergoing Mandibular Procedures
Brief Title: Study of NV-101 for Efficacy, Pharmacodynamics, and Safety in Dental Patients Undergoing Mandibular Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novalar Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NOVA 04-100
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2006-11-17 (Estimated); Status verified 2006-11

CONDITIONS: Anesthesia, Dental
Keywords: Soft Tissue Anesthesia (Numbness)
MeSH Terms: conditions — Hypesthesia | interventions — Phentolamine

INTERVENTIONS:
Drug: Phentolamine Mesylate (NV-101)

SUMMARY:
This Phase 3 study is designed as a multicenter, randomized, blinded, controlled study to evaluate the efficacy, pharmacodynamics, and safety of NV-101 administered as a submucosal injection following completion of a restorative or periodontal maintenance procedure requiring local anesthesia with an agent containing a vasoconstrictor. Local vasodilation that results in more rapid clearance of the anesthetic is the proposed mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 12 years
* Sufficiently healthy, as determined by the Investigator, to receive routine dental care
* Requires a restorative procedure in the mandible such as cavity preparation, restoration/filling, or crown or a periodontal maintenance procedure, such as teeth cleaning (non-surgical scaling and/or root planing) on the same side of the lower mouth
* Requires one or two cartridges of local anesthesia administered by one of the following intraoral injection techniques:

  * inferior alveolar nerve block;
  * Gow-Gates nerve block;
  * Vazirani-Akinosi block;
  * mental-incisive block; or
  * supraperiosteal injection.
* Dental procedure is completed within 60 minutes of the first administration of local anesthetic
* Normal lower lip and tongue sensations at baseline prior to administration of local anesthetic
* Lower lip on the side of the procedure is numb (no feeling) at the completion of the dental procedure
* Soft tissue anesthesia recovery score of zero prior to anesthetic
* Functional Assessment Battery by subject and observer rating is normal prior to anesthetic
* Negative urine pregnancy test at screening in all females of childbearing potential past menarche (includes all females except for those whose menstrual periods have not occured for greater than or equal to 1 year after menopause, who are surgically sterilized or who had a hysterectomy)
* Understands and gives written informed consent
* Subjects 12 to 17 years of age give written assent and parent(s) or legal guardian(s) give written informed consent
* Can communicate with the Investigator and study staff, and can understand and comply with the requirements of the protocol

Exclusion Criteria:

* History or presence of any condition that contraindicates routine dental care
* Requires more than two cartridges of local anesthetic (excluding supplemental injections) or use of nitrous oxide or sedatives to perform the scheduled dental procedure
* Scheduled dental procedure takes greater than 60 minutes to complete
* Unable to tolerate 1 liter of water over 5 hours
* Concurrent conditions: any incapacitating medical condition (e.g. unstable angina, uncontrolled cardiac arrhythmias, uncontrolled hypertension, uncontrolled hyperthyroidism); significant infection or inflammatory process of the oral cavity.
* Concomitant medications: use of an opioid or opioid-like analgesic (e.g. codeine, tramadol, pentazocine) within 24 hours prior to administration of anesthetic
* Allergy or intolerance to lidocaine, articaine, prilocaine, mepivacaine, epinephrine, levonordefrin, sulfites, phentolamine, or topical benzocaine
* Has used an investigational drug and/or participated in any clinical study within 30 days of study drug administration
* Has participated in this study or any previous study of phentolamine mesylate for reversal of local soft tissue anesthesia (STA)
* Any condition which, in the opinion of the Investigator, increases the risk to the subject of participating in this study or decreases the likelihood of compliance with the protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Start 2006-02; Study Completion 2006-07

PRIMARY OUTCOMES:
to determine if NV-101 accelerates time to normal sensation of the lower lip compared to control, as measured by standardized palpation procedure

SECONDARY OUTCOMES:
to determine if NV-101 accelerates the time to STAR-7 score of zero, as measured by soft tissue anesthesia questionnaire
to determine if NV-101 accelerates the time to normal function, as measured by a functional assessment battery
to determine if NV-101 accelerates the time to normal sensation of the tongue, as measured by standardized palpation procedure
to characterize the pharmacodynamic profile of NV-101, as measured by onset and offset of treatment effect
to evaluate the safety and tolerability of NV-101

CONTACTS AND LOCATIONS:
Overall Officials: Athena Papas, DMD, Principal Investigator — Tufts University
Locations (1):
- Tufts School of Dental Medicine, Boston, Massachusetts, United States